CLINICAL TRIAL: NCT04614233
Title: Targeting the Gut-brain Axis to Facilitate Weight Loss in High Fat Diet Consumers
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: PI changed institutions
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2000028769; 1R01DK126295-01A1 (NIH)
Record Dates: First submitted 2020-10-14; First posted 2020-11-03 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Overweight and Obesity
Keywords: high-fat diet consumers; gut-brain axis
MeSH Terms: conditions — Overweight; Obesity | interventions — oleoyl ethanolamine

STUDY DESIGN:
Intervention Model Description: Investigators are testing the hypotheses that high fat diet consumers will show the greatest benefit from supplementation with oleoylethanolamide (OEA) in terms of weight loss maintenance, because OEA targets brain adaptations that are related to high fat diet.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RiduZone (90% Oleoylethanolamide (OEA)) (Experimental): Participants will be randomly assigned to take 2 capsules of RiduZone (each capsule contains 90% OEA) daily for 16 months.
  Interventions: Dietary Supplement: RiduZone (90% OEA)
- Placebo (Placebo Comparator): Participants will be randomly assigned to take 2 capsules of placebo daily for 16 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: RiduZone (90% OEA) — Participants will be randomly assigned to take 2 capsules of RiduZone (each capsule contains 90% OEA ) daily for 16 months
  Arms: RiduZone (90% Oleoylethanolamide (OEA))
Drug: Placebo — Participants will be randomly assigned to take 2 capsules of placebo daily for 16 months. Placebo capsules will consist of 180mg of hypromellose.
  Arms: Placebo

SUMMARY:
The primary objective is to test if fat intake moderates the ability of oleoylethanolamide (OEA) to improve weight loss maintenance after the LEARN® weight loss program.

DETAILED DESCRIPTION:
The proposed work takes a precision medicine approach to obesity treatment and focuses specifically on weight loss maintenance. We propose to optimize a stratification strategy, using neural, metabolic and behavioral measures to identify individuals who will maintain clinically significant weight loss by daily supplementation with the fatty acid amide, oleoylethanolamide (OEA) following a gold-standard behavioral weight loss program. We will also test a model underlying the efficacy of our intervention to provide insight for the further development of therapeutic avenues. Our first aim is to conduct a randomized double-blind placebo-controlled trial to determine if fat intake moderates the ability of OEA to improve weight loss maintenance after the (LEARN®) weight loss program. We predict fat intake will strongly moderate the ability of OEA to produce clinically significant weight loss and weight loss maintenance 4- and 12-months) after LEARN and that this should not be influenced by sex.

Our second aim is to test if the Dietary Fat and Sugar intake questionnaire (DFS) is associated with measures of saturated fat intake and to optimize a clinically useful stratification strategy. Towards this end we will: (1) perform a neuroimaging study to assess brain response to a high fat milkshake (2) assess blood-based biomarkers of fat intake and synthesis; and (3) collect dietary intake records and food frequency questionnaires (FFQs). We predict that (1) the DFS predicts measures of saturated fat intake (2) that baseline dorsal striatal (DS) response to milkshake predicts weight loss in the OEA but not the placebo group and that connectome based predictive modeling (CPM) reveals a "neural fingerprint" that predicts weight loss on OEA; and (3) LASSO regression will identify baseline measures that best predict outcome to inform selection of a practical clinical stratification recommendation.

Our third aim is to test a model of OEA effectiveness. We predict that weight loss outcome is associated with shifts in fat preference and intake and these effects are mediated by increases in DS response to milkshake in the OEA but not placebo group. We will also test whether high fat diet (HFD) is associated with performance on reinforcement and cognitive measures or changes in energy expenditure or substrate utilization. If so, we will test whether these associations and their reversal by OEA contribute to outcome mediation.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-55
* Right-handed with a score of ≥ +50 on the modified Edinburgh handedness scale
* English-speaking
* BMI > 25.0
* Comfortable with the fMRI procedures during the mock scanning session and rate milkshake as at least mildly liked

Exclusion Criteria:

* Serious or unstable medical illness (e.g., cancer)
* Past or current history of alcoholism or consistent drug use
* Current major psychiatric illness as defined by DSM-IV criteria including eating disorders
* Medications that affect alertness (e.g., barbiturates, benzodiazepines, chloral hydrate, haloperidol, lithium, carbamazepine, phenytoin, etc.)
* History of major head trauma with loss of consciousness
* Ongoing pregnancy
* History of metalworking, injury with shrapnel or metal slivers, or major surgery
* History of pacemaker or neurostimulator implantation
* Known taste or smell dysfunction
* A diagnosis of diabetes
* Any known allergy to foods used in the study, or any known life-threatening food allergy
* Tobacco use

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2024-10-04 (Actual); Study Completion 2024-10-04 (Actual)

PRIMARY OUTCOMES:
Percent change in body weight | Baseline, 4 month, 8 month, and 16 months
  Weight in kg will be used to measure the percent change in body weight.
Change in absolute body weight | Baseline, 4 month, 8 month, and 16 months
  Weight in kg will be used to measure absolute body weight
Change in waist circumference | Baseline, 4 month, 8 month, 16 month
  Waist circumference to the nearest 0.1 cm
Change in hip circumference | Baseline, 4 month, 8 month, and 16 months
  Hip circumference to the nearest 0.1 cm
Change in thigh circumference | Baseline, 4 month, 8 month, and 16 months
  Thigh circumference to the nearest 0.1 cm
Change in body fat percent | Baseline, 4 month, 8 month, and 16 months
  Percentage of body fat measured with bioimpedance analysis
Change in visceral adipose tissue | Baseline, 4 month, 8 month, 16 month
  Visceral adipose tissue in liters measured with bioimpedance analysis
Change in saturated fat intake as measured by the DFS | Baseline, 4 month, 8 month, and 16 months
  Dietary fat intake will be measured monthly by diet fat and sugar intake questionnaire (DFS) and for 16 months starting from baseline. Higher scores indicate a higher frequency of saturated fat intake.
Change in saturated fat intake as measured by the ASA24 | Baseline, 4 month, 8 month, and 16 months
  Saturated fat intake will be measured monthly by the automated self-administered 24-Hour recall (ASA24) for 16 months starting from baseline.Saturated fat intake will be reported in grams.
Change in total saturated fat intake as measured by 3-day food diaries | Baseline, 4 month, 8 month, and 16 months
  Saturated fat intake will be measured monthly by 3-day food diaries for 16 months starting from baseline. The 3-day food diaries will be processed with the Nutrition Data System for Research (NDSR). Saturated fat intake will be reported in grams.
Change in total fat intake as measured by 3-day food diaries | Baseline, 4 month, 8 month, and 16 months
  Fat intake will be measured monthly by 3-day food diaries for 16 months starting from baseline. The 3-day food diaries will be processed with the Nutrition Data System for Research (NDSR). Total fat intake will be reported in grams.
Change in total saturated fat intake as measured by C-reactive protein | Baseline, 8 month
  Saturated fat intake will be measured by plasma C-reactive protein in mg/L
Change in brain response to milkshake | baseline, 8 month
  The Blood-oxygen-level-dependent response (BOLD) in the dorsal striatum to the taste of milkshake and tasteless stimuli will be measured using a 3T fMRI scanner at baseline for all participants and at month 8 for participants in the intervention group.
Change in fat perception with Visual Analogue Scale | Baseline, 4 month, 8 month, and 16 months
  Fat perception will be measured with the Visual Analogue Scale. Participants will be asked to sample Jello's and puddings of differing fat concentrations and rate their perceptual attributes at baseline, month 4, month 8, and month 16 The Visual Analogue Scale (VAS) will be used to assess perceptual attributes such as oiliness, fattiness, and creaminess, while accounting for hunger, fullness, thirst, and wanting. The VAS is a horizontal line anchored by 'not at all' at one end and 'extremely' at the other. The scale value of 'not at all' will be 0% and the scale value of 'extremely' will be 100%. Higher values indicate that a subject perceives these attributes as more intense.
Change in fat perception with General Labeled Magnitude Scale | Baseline, 4 month, 8 month, and 16 months
  Fat perception will be measured with the General Labeled Magnitude Scale (GLMS). Participants will be asked to sample Jello's and puddings of differing fat concentrations and rate their perceptual attributes at baseline, month 4, month 8, and month 16 The GLMS will assess intensity perception. The GLMS is a vertical line with quasi-logarithmic spaced labels that start at the bottom 'barely detectable' to 'strongest imaginable' at the top.
Change in fat preference with Labeled Hedonic Scale | Baseline, 4 month, 8 month, and 16 months
  Fat preference will be measured. Participants will be asked to sample Jello's and puddings of differing fat concentrations and rate their hedonic attributes at baseline, month 4, month 8, and month 16 The Labeled Hedonic Scale (LHS) will assess liking. The LHS is a vertical line with quasi-logarithmic spaced labels that start at the bottom with 'most imaginable dislike' and go to 'most imaginable like' at the top, with the label 'neutral' in the middle. The scale value of 'most imaginable dislike' will be -100; the scale value of 'neutral' will be 0; the scale value of 'most imaginable like' will be 100. Higher values indicate greater liking of the sample.
Change in sensitivity to the long-chain oleic acid C18:1 - measured by a 3-alternative forced choice test | Baseline, 4 month, 8 month, 16 month
  Subjects will be presented with a set of three samples, one test sample with a specific concentration of fat and two control samples. Subjects will be instructed to choose "the odd one out". If the subject chooses incorrectly, the fat concentration of the fatty test sample will be increased in the next set of three samples. If the subject chooses correctly, the next set of three samples will have the fatty test sample would contain the same fat concentration as in the previously correctly identified set with two control samples. This will continue until the subject correctly chooses the fatty test sample three times consecutively.
Change in sugar perception with General Labeled Magnitude Scale | Baseline, 4 month, 8 month, and 16 months
  Sugar perception will be measured with the General Labeled Magnitude Scale. Participants will be asked to sample Jello's and puddings of differing sugar concentrations and rate their perceptual and attributes at baseline, month 4, month 8 , and month 16 The GLMS will assess intensity perception. The GLMS is a vertical line with quasi-logarithmic spaced labels that start at the bottom 'barely detectable' to 'strongest imaginable' at the top.
Change in sugar preference with Labeled Hedonic Scale | Baseline, 4 month, 8 month, and 16 months
  Sugar perception will be measured with the Labeled Hedonic Scale. Participants will be asked to sample Jello's and puddings of differing sugar concentrations and rate their hedonic attributes at baseline, month 4, month 8, and month 16 The LHS will assess liking. The LHS is a vertical line with quasi-logarithmic spaced labels that start at the bottom with 'most imaginable dislike' and go to 'most imaginable like' at the top, with the label 'neutral' in the middle.
Change in fat concentration preference measured by the Monell forced choice test | Baseline, 4 month, 8 month, and 16 months
  Fat concentration preference will be measured by the Monell forced-choice test. Participants will be asked to sample Jello's and puddings of differing fat concentrations at baseline, month 4, month 8 , and month 16.
  Subjects will be presented with pairs of puddings of varying fat concentrations in a two-series test. Subjects will taste two puddings of different fat concentrations and indicate their preferred pudding. The following pairs of puddings will be presented based on the subject's previous choice. This will continue until selection of the same fat concentration twice relative to both a lower and a higher concentration, or until the lowest or highest concentration is chosen twice consecutively.
Change in sweet concentration preference measured by the Monell forced choice test | Baseline, 4 month, 8 month, and 16 months
  Sweet concentration preference will be measured by the Monell forced-choice test. Participants will be asked to sample Jello's and puddings of differing sugar concentrations at baseline, month 4, month 8 , and month 16.
  Subjects will be presented with pairs of puddings/Jello's of varying sugar concentrations in a two-series test. Subjects will taste two puddings/Jello's of different sugar concentrations and indicate their preference. The following pairs of puddings/Jello's will be presented based on the subject's previous choice. This will continue until selection of the same sugar concentration twice relative to both a lower and a higher concentration, or until the lowest or highest concentration is chosen twice consecutively.
Change in food reinforcement with RED-13 | Baseline and 8 month
  The relative reinforcing value of foods will be measured using the Reward-Related Eating (RED-13) Questionnaire. This questionnaire results in a score from 0 as the lowest measure of reward-based eating drive and 36 as the highest.
Change in food reinforcement with Becker DeGroot Markov Auction Task | Baseline and 8 month
  The relative reinforcing value of foods will be measured using a computerized auction task at baseline and month 8. The relative reinforcing value of foods will be measured with a modified version of the Becker DeGroot Markov Auction task. The outcome measure is willingness to pay, such that higher willingness to pay indicates higher relative reinforcing value of foods.
Change in cognition with Kirby Delay Discounting | Baseline, 4 month, 8 month, and 16 months
  A neuropsychological test battery will be performed to assess obesity or dopamine-related differences in cognition at baseline, month 4, month 8, and month 16. The neuropsychological test battery will include Kirby Delay Discounting, which measures temporal discounting (tendency for people to prefer small, immediate, monetary rewards over larger, delayed rewards). The steepness of the discounting curve represents the tendency for temporal discounting, such that a more steeply declining curve indicates a tendency to devalue rewards as they become more temporally remote.
Change in cognition with the Relational Task | Baseline, 4 month, 8 month, and 16 months
  A neuropsychological test battery will be performed to assess obesity or dopamine-related differences in cognition at baseline, month 4, month 8, and month 16. The neuropsychological test battery will include the Relational Task which measures visual relational processing. The number of correct responses in the relational condition is the outcome measurement, such that more correct responses indicates higher visual relational processing.
Change in cognition with Penn Progressive Matrices Test | Baseline, 4 month, 8 month, and 16 months
  A neuropsychological test battery will be performed to assess obesity or dopamine-related differences in cognition at baseline, month 4, month 8, and month 16. The neuropsychological test battery will include the Penn Progressive Matrices Test, which measures fluid intelligence. The number of correct responses is the outcome measurement, such that more correct responses indicates higher fluid intelligence.
Change in cognition with Oral Reading Recognition Test | Baseline, 4 month, 8 month, and 16 months
  A neuropsychological test battery will be performed to assess obesity or dopamine-related differences in cognition at baseline, month 4, month 8, and month 16. The neuropsychological test battery will include the Oral Reading Recognition Test, which measures language decoding and reading. The score based on accuracy is the outcome measure, such that a higher score indicates higher language decoding and reading ability.
Change in cognition with Variable Short Penn Line Orientation Test | Baseline, 4 month, 8 month, and 16 months
  A neuropsychological test battery will be performed to assess obesity or dopamine-related differences in cognition at baseline, month 4, month 8, and month 16. The neuropsychological test battery will include the Variable Short Penn Line Orientation Test, which measures visuospatial processing. The number of correct responses is the outcome measure, such that a higher number of correct responses indicates higher visuospatial processing ability.
Change in cognition with Matrix Reasoning Task (Core NMOB) | Baseline, 4 month, 8 month, and 16 months
  A neuropsychological test battery will be performed to assess obesity or dopamine-related differences in cognition at baseline, month 4, month 8, and month 16. The neuropsychological test battery will include the Core Neuropsychological Measures for Obesity and Diabetes (Core NMOB). Core NMOB includes the Matrix Reasoning task, which reflects general cognitive ability or nonverbal reasoning ability. Accuracy across 35 trials is the outcome measure, such that higher accuracy indicates higher general cognitive ability or nonverbal reasoning ability.
Change in cognition with Digit Symbol Substitution (Core NMOB) | Baseline, 4 month, 8 month, and 16 months
  A neuropsychological test battery will be performed to assess obesity or dopamine-related differences in cognition at baseline, month 4, month 8, and month 16. The neuropsychological test battery will include the Core Neuropsychological Measures for Obesity and Diabetes (Core NMOB). Core NMOB includes the Digit Symbol Substitution task, which reflects processing speed. The number of correctly matched symbols, within the administration time (90 seconds) is the outcome measure, such that higher number of correctly matched symbols indicates higher processing speed.
Change in cognition with Go/No-Go Task (Core NMOB) | Baseline, 4 month, 8 month, and 16 months
  A neuropsychological test battery will be performed to assess obesity or dopamine-related differences in cognition at baseline, month 4, month 8, and month 16. The neuropsychological test battery will include the Core Neuropsychological Measures for Obesity and Diabetes (Core NMOB). Core NMOB includes the Go/No-Go task, which reflects response inhibition. The sensitivity index (d') and commission error rate is the outcome measure, such that higher d' and lower commission error rates indicate higher response inhibition.
Change in cognition with Penn Word Memory Test | Baseline, 4 month, 8 month, and 16 months
  A neuropsychological test battery will be performed to assess obesity or dopamine-related differences in cognition at baseline, month 4, month 8, and month 16. The neuropsychological test battery will include the Penn Word Memory Test, which measures verbal episodic memory. The number of correct responses is the outcome measure, such that a higher number of correct responses indicates higher verbal episodic memory.
Change in cognition with Dimensional Change Card Sorting (Core NMOB) | Baseline, 4 month, 8 month, and 16 months
  A neuropsychological test battery will be performed to assess obesity or dopamine-related differences in cognition at baseline, month 4, month 8, and month 16. The neuropsychological test battery will include the Core Neuropsychological Measures for Obesity and Diabetes (Core NMOB). Core NMOB includes the Dimensional Change Card Sorting task, which reflects cognitive flexibility and task-switching ability. The accuracy score is the outcome measure, such that higher accuracy indicates higher cognitive flexibility and task-switching ability.
Change in cognition with Picture Sequence Memory (Core NMOB) | Baseline, 4 month, 8 month, and 16 months
  A neuropsychological test battery will be performed to assess obesity or dopamine-related differences in cognition at baseline, month 4, month 8, and month 16. The neuropsychological test battery will include the Core Neuropsychological Measures for Obesity and Diabetes (Core NMOB). Core NMOB includes the Picture Sequence Memory task, which reflects learning and memory. The accuracy score is the outcome measure, such that higher accuracy indicates higher learning and memory abilities.
Change in cognition with Stockings of Cambridge (SOC) test (CANTAB) | Baseline, 4 month, 8 month, and 16 months
  A neuropsychological test battery will be performed to assess obesity or dopamine-related differences in cognition at baseline, month 4, month 8, and month 16. The neuropsychological test battery will include the Cambridge Neuropsychological Test Automated Battery (CANTAB). The CANTAB includes the Stockings of Cambridge test, which reflects spatial planning. Outcome measures assess the problem difficulty level reached, mean moves used and thinking time are the outcome measures. Scores will be compared to normative data from age and sex-matched peers.
Change in cognition with Intra-Extra Dimensional Set Shift test (CANTAB) | Baseline, 4 month, 8 month, and 16 months
  A neuropsychological test battery will be performed to assess obesity or dopamine-related differences in cognition at baseline, month 4, month 8, and month 16. The neuropsychological test battery will include the Cambridge Neuropsychological Test Automated Battery (CANTAB). The CANTAB includes the Intra-Extra Dimensional Set Shift test, which reflects rule acquisition and reversal. Outcome measures assess the number of errors made, the number of trials completed, the number of stages completed and latency. Scores will be compared to normative data from age and sex-matched peers.
Change in cognition with delayed non-matching to sample test (CANTAB) | Baseline, 4 month, 8 month, and 16 months
  A neuropsychological test battery will be performed to assess obesity or dopamine-related differences in cognition at baseline, month 4, month 8, and month 16. The neuropsychological test battery will include the Cambridge Neuropsychological Test Automated Battery (CANTAB). The CANTAB includes the delayed non-matching to sample test, which reflects visuospatial memory. Outcome measures include latency (the participant's speed of response), the number of correct patterns selected and a statistical measure giving the probability of an error after a correct or incorrect response. Scores will be compared to normative data from age and sex-matched peers.
Change in cognition with Paired Associates Learning task (CANTAB) | Baseline, 4 month, 8 month, and 16 months
  A neuropsychological test battery will be performed to assess obesity or dopamine-related differences in cognition at baseline, month 4, month 8, and month 16. The neuropsychological test battery will include the Cambridge Neuropsychological Test Automated Battery (CANTAB). The CANTAB includes the Paired Associates Learning task, which assesses episodic memory and new learning. Outcome measures include the errors made by the participant, the number of trials required to locate the pattern(s) correctly, memory scores and stages completed. Scores will be compared to normative data from age and sex-matched peers.
Change in cognition with Probabilistic-Feedback Reward Task | Baseline, 4 month, 8 month, and 16 months
  A neuropsychological test battery will be performed to assess obesity or dopamine-related differences in cognition at baseline, month 4, month 8, and month 16. The neuropsychological test battery will include the Probabilistic-Feedback Reward Task, which assesses the ability to learn from positive and negative outcome. Outcome measures include the number of times a symbol associated with positive feedback is chosen and the number of times a symbol associated with negative feedback is avoided. Scores will be compared to normative data from age and sex-matched peers.
Change in resting energy expenditure | Baseline and 8 month
  Indirect Calorimetry (IC) will be performed to measure fasting resting energy expenditure at baseline and month 8.
Change in respiratory exchange ratio | Baseline and 8 month
  Indirect Calorimetry (IC) will be performed to measure fasting respiratory exchange ratio at baseline and month 8

SECONDARY OUTCOMES:
Change in Healthy Eating Index (HEI) | Baseline, 4 month, 8 month, 16 month
  The overall Healthy Eating Index 2015 (HEI-2015) score will be calculated for each participant from 3-day food diaries processed through NDSR. This score is made up of 13 components that reflect recommendations in the 2015-2020 Dietary Guidelines for Americans. The maximum score for the HEI is 100, where points are awarded based on adequate intakes of total fruit, whole fruits, total vegetables, greens and beans, whole grains, dairy, protein foods, seafood and plant proteins, and unsaturated fatty acids. Points are also awarded for moderate intakes of refined grains, sodium, added sugars and saturated fats.
Change in 3-day food diary total solid fat intake | Baseline, 4 month, 8 month, 16 month
  Solid fat intake will be measured monthly by 3-day food diaries for 16 months starting from baseline. The 3-day food diaries will be processed with the Nutrition Data System for Research (NDSR) and solid fat intake will be reported in grams.
Change in saturated fat intake measured by plasma cholesterol | Baseline, 8 month
  Plasma cholesterol LDL/HDL will be measured at baseline and month 8
Change in saturated fat intake measured by plasma triglycerides | Baseline, 8 month
  Plasma triglycerides will be measured at baseline and month 8

CONTACTS AND LOCATIONS:
Locations (1):
- Modern Diet and Physiology Research Lab, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Fang X, Davis X, Flack KD, Duncan C, Li F, White M, Grilo C, Small DM. Dietary adaptation for weight loss maintenance at Yale (DAWLY): Protocol and predictions for a randomized controlled trial. Front Nutr. 2022 Jul 28;9:940064. doi: 10.3389/fnut.2022.940064. eCollection 2022. PMID 35967820

DOCUMENTS (1):
  • Informed Consent Form (2023-11-20): https://cdn.clinicaltrials.gov/large-docs/33/NCT04614233/ICF_000.pdf